CLINICAL TRIAL: NCT05922111
Title: Comparison of Labor Induction With Cervical Ripening Balloon, One Versus Tweleve Hours Placement: a Randomized Controlled Trial
Brief Title: Cervical Ripening Balloon for 12 Hours vs. 1 Hour.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0602-21-RMB CTIL
Record Dates: First submitted 2022-11-27; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Induction of Labor

STUDY DESIGN:
Intervention Model Description: This will be an open-label,1:1, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical ripening balloon for 1 hour (Experimental): Eligible women will undergo the usual procedure of CRB insertion using a double lumen Cook cervical ripening balloon (CCRB). The CRB will be removed approximately after an hour in the intervention group and thereafter, the women will proceed amniotomy or Pitocin use at the discretion of the labor and delivery physician
  Interventions: Device: cervical ripening balloon for one hour
- cervical ripening balloon for 12 hours (Active Comparator): Eligible women will undergo the usual procedure of CRB insertion using a double lumen Cook cervical ripening balloon (CCRB). The CRB will be removed approximately after 12 hours in the control group and thereafter, the women will proceed amniotomy or Pitocin use at the discretion of the labor and delivery physician
  Interventions: Device: cervical ripening balloon for twelve hours

INTERVENTIONS:
Device: cervical ripening balloon for one hour — The cervical ripening balloon will be left in place for one hour and after balloon removal the induction of labor will proceed at the discretion of the attending physician at labor and delivery room
  Arms: cervical ripening balloon for 1 hour
Device: cervical ripening balloon for twelve hours — The cervical ripening balloon will be left in place for for twelve hours and after balloon removal the induction of labor will proceed at the discretion of the attending physician at labor and delivery room
  Arms: cervical ripening balloon for 12 hours

SUMMARY:
The aim of this study is a comparison of induction of labor with a cervical ripening balloon left in place for one hour compared to twelve hours. The primary outcome is time to delivery.

Women admitted for induction of labor will be recruited and randomized to either a cervical ripening balloon for one hour or twelve hours. the management of delivery after the extraction of the balloon will be left to the discretion of the attending physician.

DETAILED DESCRIPTION:
The common IOL techniques used for pregnant women with unfavorable cervix might be specified to either mechanical induction via cervical ripening balloon (CRB) or pharmacological induction. The insertion of a CRB is believed to mechanically ripen the uterine cervix with a better safety profile than prostaglandins. The duration of the balloon placement varied considerably, and it was commonly placed for 12-24 hours. Nevertheless, recent randomized controlled studies have demonstrated favorable results following only 6 hours of CRB placement with or without additional administration of oxytocin. We believe that mechanical ripening of the cervix can be achieved even less than six hours. Our study aims to evaluate the time to delivery and pregnancy outcomes after placement of CRB of only 1 hour compared to either 6 or 12 hours.

Study Protocol:

1. Women planned for induction of labor will be approached by a trained resident and will sign informed consent.
2. All participants will be randomized to either one hour or twelve hours CRB placement using a computer program randomization scheme, block size of 20, by the department research coordinator who will keep the sequential in sealed envelopes.
3. Demographic parameters will be retrieved from the computerized database of Rambam Medical Center (RMC).
4. Eligible women will undergo the usual procedure of CRB insertion using a double lumen Cook cervical ripening balloon (CCRB). The CRB will be removed approximately after an hour in the intervention group and after twelve hours in the control group. Thereafter, the women will proceed amniotomy or Pitocin use at the discretion of the labor and delivery physician

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous or multiparous gravidas
2. Gestational age ≥ 370/7 to 416/7 gestational weeks
3. Age 18-45
4. Signed informed consent

Exclusion Criteria:

1. Contraindications for vaginal delivery
2. Multifetal gestation
3. Rupture of membranes
4. Bishop score > 6
5. The cervix is dilated to more than 2 cm
6. Previous caesarean delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
insertion to delivery time interval | From date of balloon insertion until the date of delivery, assessed up to 4 days
  The time interval between balloon insertion to delivery

SECONDARY OUTCOMES:
to compare the mode of delivery | From date of balloon insertion until the date of delivery, assessed up to 4 days
  Mode of delivery
to compare the time to active and second stage of labor | From date of balloon insertion until the date of delivery, assessed up to 4 days
  Time to active and second stage of labor
to compare the rate of chorioamnionitis | From date of balloon insertion until the date of discharge, assessed up to 8 days
  Rate of chorioamnionitis
to compare the rate of post-partum hemorrhage | From date of balloon insertion until the date of discharge, assessed up to 8 days
  Rate of post-partum hemorrhage and need for blood transfusion
to compare the need for blood transfusion | From date of balloon insertion until the date of discharge, assessed up to 8 days
  the need for blood transfusion
to compare the rate of anal sphincter injuries | From date of balloon insertion until the date of discharge, assessed up to 8 days
  Rate of obstetric anal sphincter injuries
To compare the length of maternal hospital stay | From date of balloon insertion until the date of discharge, assessed up to 8 days
  Length of maternal hospital stay
To compare the overall satisfaction rate | From date of balloon insertion until the date of discharge, assessed up to 8 days
  Overall satisfaction using the Birth satisfaction scale questionnaire with higher score means a better outcome. minimal score 30, maximal score 150.
To compare the Apgar score between the groups | at the date of delivery
  Apgar score - higher score means better outcome. Minimal score is 0, maximal Apgar score is 10.
To compare the rate of neonatal acidemia between the groups | From date of delivery until the date of neonate discharge, assessed up to 14 days
  Neonatal acidemia
To compare the rate of admission to neonatal intensive care unit between the groups | From date of delivery until the date of neonate discharge, assessed up to 14 days
  Admission to neonatal intensive care unit
To compare the rate of Respiratory complications between the groups | From date of delivery until the date of neonate discharge, assessed up to 14 days
  Respiratory complications
To compare the rate of neonatal sepsis between the groups | From date of delivery until the date of neonate discharge, assessed up to 14 days
  Neonatal sepsis
To compare the rate of birthweightbetween the groups | at the date of delivery
  Birthweight in grams

CONTACTS AND LOCATIONS:
Overall Officials: Naphtali Justman, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No
Study protocol and informed consent form will be shared upon request from the corresponding author